CLINICAL TRIAL: NCT05797311
Title: The Effect of Proprioceptive Neuromuscular Facilitation and Shoulder Stabilization Exercises on Pain, Quality of Life and Functionality in Adhesive Capsulitis Treatment
Brief Title: The Effect of PNF and Shoulder Stabilization Exercises on Pain, QoL and Functionality in Patient With AC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, osman coban, Principal Investigator, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UskudarUniversity
Record Dates: First submitted 2023-03-10; First posted 2023-04-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive Capsulitis; pain; Proprioceptive Neuromuscular Facilitation; Shoulder Stabilization Exercises
MeSH Terms: conditions — Bursitis; Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Group (Experimental): After classical physiotherapy consisting of 40 minutes of hot pack, TENS, US and Exercise (a set of stretching exercises including Wand and Codman pendulum exercises) was applied by an experienced Physiotherapist, additional PNF exercises were performed once a day, 5 times a week by the same Physiotherapist in the cases in the PNF group. It will be applied for a total of 3 weeks (Total of 15 sessions).
  1. PNF contract-relax to subscapularis and internal rotators (7 Sec of contraction and 15 Sec of relaxation in external rotation, 5 repetitions) Followed by facilitation of D2 Flexion patterns for 5 repetitions.
  2. PNF all scapular patterns with Rhythmic initiation and repeated contractions Technique .
  Interventions: Other: Proprioceptive Neuromuscular Facilitation (PNF)
- Stabilization Group (Other): After classical physiotherapy consisting of 40 minutes of hot pack, TENS, US and Exercise (a set of stretching exercises including Wand and Codman pendulum exercises) was applied by an experienced Physiotherapist, stabilization exercises were performed by the same Physiotherapist once a day, 5 times a week, for a total of 5 times a week. It will be applied for 3 weeks (Total of 15 sessions).
  1. scapular stabilization exercises
  2. stabilization exercise for the shoulder joints.
  In all the exercises, the subjects maintained the position for 10 seconds, and they took a rest for 3 seconds. Ten repetitions was considered one set, and the subjects conducted three sets. A break of 3 minutes was given between each set.
  Interventions: Other: Shoulder Stabilization Exercises

INTERVENTIONS:
Other: Proprioceptive Neuromuscular Facilitation (PNF) — Proprioceptive Neuromuscular Facilitation (PNF) techniques are a therapeutic exercise approach developed based on functional activities in daily life. At the stage of regaining movement and function, it creates models similar to functional activities.
  Arms: PNF Group
Other: Shoulder Stabilization Exercises — Scapular stabilization exercise and stabilization exercise for the shoulder joints
  Arms: Stabilization Group

SUMMARY:
Adhesive capsulitis (AC), also known as frozen shoulder, is an insidious, painful condition of the shoulder lasting more than 3 months. This inflammatory condition causing fibrosis of the glenohumeral joint capsule is accompanied by gradual progressive stiffness and marked limitation of range of motion (typically external rotation). Patients experiencing this condition often suffer from poor quality of life due to the limitation of both the active and passive range of shoulder mobility. The prevalence of frozen shoulder is between 2-5% and is more common in women. Along with the increase in comorbidities and changes in lifestyle, the incidence of FS is increasing. However, the natural history and pathogenesis of adhesive capsulitis have not been widely studied and are still unknown. Adhesive capsulitis presents clinically as shoulder pain with progressive restricted movement, both active and passive, with normal radiographic scans of the glenohumeral joint. Classically, it progresses prognostically with 3 overlapping stages: pain (stage 1, lasting 2-9 months), stiffness (stage 2, lasting 4-12 months), and healing (stage 3, lasting 5-24 months). However, this is an estimated time frame and many patients may still experience symptoms after 6 years. Treatment modalities include conservative (ie, steroid injection, physiotherapy) and operative (ie, distension arthrography, manipulation under anesthesia, and arthroscopic release).

Various physical therapy treatments commonly used in the treatment of adhesive capsulitis include ice pack, hot pack, transcutaneous electrical nerve stimulation and active and passive ROM exercises, joint mobilization techniques, proprioceptive neuromuscular facilitation (PNF), supervised home exercise programs, and Kinesio taping.

DETAILED DESCRIPTION:
There are studies on the application of PNF techniques in proprioceptive neuromuscular facilitation (PNF), sports injuries, orthopedics, cardiorespiratory and neurological conditions developed by Knott and Kabat. Recently, the application of these techniques in orthopedic conditions has been developing. However, studies have been conducted to find out the effect of PNF therapy on Adhesive Capsulitis, but there is conflicting evidence between them. Although some studies have suggested PNF, determining which technique is better in the treatment of AC remains controversial and needs to be answered. Therefore, in our study, it was aimed to compare the effects and advantages of proprioceptive neuromuscular exercises and shoulder stabilization exercises applied in the treatment of patients with Adhesive capsulitis and to evaluate the acute effects of these exercises on shoulder movements.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20- 65 years diagnosed with unilateral Stage II adhesive capsulitis by magnetic resonance imaging
* Shoulder pain persisting for at least 3 months
* VAS pain score equal to or greater than 5/10
* Patients who agreed to participate in the study

Exclusion Criteria:

* - Receiving physical therapy or manual therapy on the same shoulder within 1 year
* Having mental and cognitive problems,
* Patients who have undergone surgical procedure/injection/manipulation to the shoulder joint for any reason
* Neurological disorders that affect shoulder function during daily activities
* Pain or discomfort in the cervical spine, elbow, wrist, or hand
* Other pathological conditions concerning the shoulder (rotator cuff tear, tendinitis, etc.)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Evaluation | Change from baseline to week 3
  The Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line, and the patient is asked to draw a line on this line to indicate where his condition is appropriate.

SECONDARY OUTCOMES:
Manual Muscle Testing | Change from baseline to week 3
  During the testing of muscle strength without using any device ("manual muscle testing"), the evaluation system (Medical Research Council (MRC)) scale, which is widely used all over the world, is used. It is the evaluation of motion in the context of gravity.
Joint Range of Motion | Change from baseline to week 3
  A Goniometer is the most common tool for measuring range of motion of the joints of the body. It uses a stationary arm, fulcrum, and movement arm to measure joint angles from the axis of the joint. Making a ROM measurement by using a goniometer requires training for reliable results. See the goniometry collection of pages for instructions on how to correctly (reliably and accurately) place the goniometer when measuring range of motion.
DASH (Arm, Shoulder and Hand Problems Questionnaire) | Change from baseline to week 3
  The DASH questionnaire consists of 3 parts. The first part consists of 30 questions. 21 questions evaluate the degree of difficulty of the patient in daily activities, 5 questions evaluate the symptomatic features of pain, and 4 questions evaluate social function, self-confidence and sleep.
Short Form 12 (SF-12) | Change from baseline to week 3
  SF-12, a measure of Health-Related Quality of Life, can be used in age, disease and treatment groups. It is a shortened version of the SF-36 and contains 12 questions, each with two to five answer options. The patient is told to choose the option that best suits him/her. The SF-12 covers eight dimensions: general health, physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. A physical and mental health score, each ranging from 0 to 100, can be calculated using scoring algorithms. Scores are calibrated to a mean score of 50, or the norm, with lower scores representing worse and higher scores representing better Health-Related Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: safiye gul abat, PT, Principal Investigator — Uskudar University
Locations (1):
- Uskudar University Health Science, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho CH, Bae KC, Kim DH. Treatment Strategy for Frozen Shoulder. Clin Orthop Surg. 2019 Sep;11(3):249-257. doi: 10.4055/cios.2019.11.3.249. Epub 2019 Aug 12. PMID 31475043
- [Background] Cho CH, Song KS, Kim BS, Kim DH, Lho YM. Biological Aspect of Pathophysiology for Frozen Shoulder. Biomed Res Int. 2018 May 24;2018:7274517. doi: 10.1155/2018/7274517. eCollection 2018. PMID 29992159
- [Background] Challoumas D, Biddle M, McLean M, Millar NL. Comparison of Treatments for Frozen Shoulder: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Dec 1;3(12):e2029581. doi: 10.1001/jamanetworkopen.2020.29581. PMID 33326025
- [Background] Barbosa F, Swamy G, Salem H, Creswell T, Espag M, Tambe A, Clark D. Chronic adhesive capsulitis (Frozen shoulder): Comparative outcomes of treatment in patients with diabetes and obesity. J Clin Orthop Trauma. 2019 Mar-Apr;10(2):265-268. doi: 10.1016/j.jcot.2018.02.015. Epub 2018 Feb 25. PMID 30828190
- [Background] Kraal T, Visser C, Sierevelt I, Beimers L. How to treat a frozen shoulder? A survey among shoulder specialists in the Netherlands and Belgium. Acta Orthop Belg. 2016 Mar;82(1):78-84. PMID 26984658
- [Background] Neviaser AS, Hannafin JA. Adhesive capsulitis: a review of current treatment. Am J Sports Med. 2010 Nov;38(11):2346-56. doi: 10.1177/0363546509348048. Epub 2010 Jan 28. PMID 20110457
- [Background] Tedla JS, Sangadala DR. Proprioceptive neuromuscular facilitation techniques in adhesive capsulitis: a systematic review and meta-analysis. J Musculoskelet Neuronal Interact. 2019 Dec 1;19(4):482-491. PMID 31789299
- [Background] Balci NC, Yuruk ZO, Zeybek A, Gulsen M, Tekindal MA. Acute effect of scapular proprioceptive neuromuscular facilitation (PNF) techniques and classic exercises in adhesive capsulitis: a randomized controlled trial. J Phys Ther Sci. 2016 Apr;28(4):1219-27. doi: 10.1589/jpts.28.1219. Epub 2016 Apr 28. PMID 27190456
- [Background] Park SI, Choi YK, Lee JH, Kim YM. Effects of shoulder stabilization exercise on pain and functional recovery of shoulder impingement syndrome patients. J Phys Ther Sci. 2013 Nov;25(11):1359-62. doi: 10.1589/jpts.25.1359. Epub 2013 Dec 11. PMID 24396188
- [Background] Mezian K, Coffey R, Chang KV. Frozen Shoulder(Archived). 2023 Aug 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482162/ PMID 29489251